CLINICAL TRIAL: NCT04394572
Title: Identification of New Diagnostic Protein Markers for Colorectal Cancer in Circulating Tumor Exosomes
Brief Title: Identification of New Diagnostic Protein Markers for Colorectal Cancer
Acronym: EXOSCOL01
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19143*
Record Dates: First submitted 2020-01-31; First posted 2020-05-19 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: exosome ; colon cancer; integrin; matrix metalloproteinases
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal cancer: Patients with and without colorectal cancer
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — All patients included in the study will have blood sample

SUMMARY:
The search for biochemical markers in patient's blood for non-invasive colorectal cancer diagnostic has not yielded satisfactory results to date. The search for blood in the stool by enzymatic techniques has certainly allowed the diminution of colorectal cancer mortality but its low sensitivity is still a disadvantage. The new immunological tests for search blood test in the stool are more sensitive and more specific but still insufficient. The originality of this project is based on the use of new technology developed in fundamental research based on the detection of circulating exosomes from tumor cells in the patient's serum. The detection of protein markers transported by tumor exosomes is original and innovative approach because it's still not considered in the literature. The use of innovative and non-invasive health technologies for the patient is an important factor in the care of patients in their health care journey. The non-invasive nature of the project could reduce the reticence of patients to participate in cancer screening.

The results expected from the study can have a direct impact on the management of patients suspected of having colon cancer and thus make it possible to optimize the earliness of their diagnosis.

DETAILED DESCRIPTION:
In terms of frequency, colorectal cancer is the third most common cancer diagnosed in men and the second in women. Screening for colon and rectal cancer is based on the search for blood in the stool. The detection of occult bleeding is an indication for colonoscopy to find the origin of this bleeding. In this context, the search for biochemical markers in the blood of patients for diagnostic purposes has not yielded satisfactory results to date. Cancer cells, including colorectal cancer cells, release extracellular vesicles that contain proteins, mRNAs, DNA that can be transferred to neighboring cells but that also circulate through the blood stream and can modulate tumor progression and metastatic spread. These extracellular vesicles are of two types: exosomes (40 to 100 nm in diameter) formed by budding of endosome membranes and microvesicles (100 to 1000 nm in diameter) resulting from the budding of plasma membrane. Exosomes carry transmembrane proteins on their surface, called tetraspanins (CD9, CD63, CD81) but they also contain proteases involved in the degradation of the extracellular matrix, integrins involved in the tropism of metastases, and matrix macromolecules involved in the control of tumor invasion. The working hypothesis is that some of these exosomal proteins may be good diagnostic and / or prognostic markers for colorectal cancer. This project will aim to isolate exosomes from patient blood and to quantify previously cited proteins according to the accreditation criteria of clinical laboratory biology analyzes. For this purpose, exosomes will be isolated from sera of patients and their number, size and protein composition will be characterized. This project is an innovative and non-invasive prospective approach in the screening of protein markers for colorectal cancer diagnostic and / or prognostic.

ELIGIBILITY:
Inclusion Criteria:

* Immunoassay for stool positive blood test or family screening
* Patients seen in consultation for a colonoscopy
* Patient who gave their consent for the study (signed consent form)
* Patient affiliated to a health insurance plan

Exclusion Criteria:

* History of other cancers (except for cervical cancer or basal cell carcinoma treated for curative purposes)
* Patient under chemotherapy
* Patients with a known familial mutation (APC, MSI, MYH)
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic performances of markers derived from circulating tumor exosomes in the context of colorectal cancer, focusing on macromolecules | Day 1
  Sensitivity and specificity of macromolecules
Diagnostic performances of markers derived from circulating tumor exosomes in the context of colorectal cancer, focusing on integrins | Day 1
  Sensitivity and specificity of integrins
Diagnostic performances of markers derived from circulating tumor exosomes in the context of colorectal cancer, focusing on metallo proteases | Day 1
  Sensitivity and specificity of metallo proteases

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided